CLINICAL TRIAL: NCT03109028
Title: Stepped Care Model Supporting Mental Health in Refugees and Asylum Seekers
Brief Title: Mental Health in Refugees and Asylum Seekers
Acronym: MEHIRA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: Zentralinstitut für Seelische Gesundheit Mannheim (Other); University of Potsdam (Other); University of Ulm (Other); Philipps University Marburg (Other); RWTH Aachen University (Other); Ludwig-Maximilians - University of Munich (Other)
Responsible Party: Principal Investigator, Malek Bajbouj, Prof. Dr. med., Charite University, Berlin, Germany
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 01VSF16061
Record Dates: First submitted 2017-04-06; First posted 2017-04-11 (Actual); Last update posted 2022-02-18 (Actual); Status verified 2022-02

CONDITIONS: Affective Disorders
MeSH Terms: conditions — Mood Disorders | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment as Usual (Active Comparator): Regular standard psychiatric health care including all feasible interventions including medication, psychotherapy and social work.
  Interventions: Other: Treatment as Ususal
- Stepped and Collaborative Care Modell (Experimental): A stepped and collaborative treatment model with varying stepped psychotherapeutic interventions for adult and adolescent refugees.
  Interventions: Behavioral: Peer-to-Peer-Groupintervention; Behavioral: Smartphone-based-Intervention; Behavioral: Gendersensitive-Groupintervention; Behavioral: Empowerment-Groupintervention; Behavioral: Adolescent-Groupintervention

INTERVENTIONS:
Behavioral: Peer-to-Peer-Groupintervention — Target group: Adult participants with mild to moderate depressive symptoms who prefer therapists with the same cultural background.
  Therapists: Recruitment of psychosocial counselors within refugee community who have sufficient German or English language knowledge. Counselors will be trained for a time period of two months.
  Content: Vulnerability and resilience factors; Self-efficacy strategies; Causes and consequences of stress; Possibilities on accelerating the integration process; Strategies preventing violence and radicalization Form of therapy: Group-based intervention for a time period of three months; Two times per week with each session enduring 90 minutes; Group size between 8-10 participants; Headed by two psychosocial counselors.
  Arms: Stepped and Collaborative Care Modell
Behavioral: Smartphone-based-Intervention — Target group: Participants with moderate depressive symptoms who prefer an internet-based intervention.
  Content: Five modules with 20 exercises elaborating on psycho-education, treatment options, self-management and diagnostics.
  Form of therapy: Participants receive regular emails and sms to encourage steady participation via the internet-based smartphone-application. Weekly questionnaires ascertain the degree of participants symptomatology.
  Arms: Stepped and Collaborative Care Modell
Behavioral: Gendersensitive-Groupintervention — Target group: Vulnerable group of adult women while taking cultural characteristics into account Therapists: Recruitment of psychosocial counselors (similar to Peer-to-Peer-Intervention); Training and supervision of gender-specific aspects.
  Content: Focus on psycho-education which consider women specific topics such as gender-differences in symptoms and prevalence in psychic stress related and trauma disorders; physical, psychic and psychosocial consequences of traumatic and violent experiences; gender-specific risk and safety factors; stress and emotional self-regulation Form of therapy: Group-based intervention for a time period of three months; Two times per week with each session enduring 90 minutes; Group size between 8-10 participants; Headed by two female psychosocial counselors.
  Arms: Stepped and Collaborative Care Modell
Behavioral: Empowerment-Groupintervention — Target group: Gender-sensitive group with mild to moderate depressive symptoms. Therapists: Psychologists and doctors in psychotherapeutic advanced training; The therapist-training lasts for three months with continued supervision during the intervention.
  Content: Low-threshold intervention based on the treatment of depression; psycho-education about psychic burdens, trauma, stress and grief as well as vulnerability and resilience factors; Problem solving and self-actualization strategies.
  Form of therapy: Group-based intervention for a time period of two months; Two times per week with each session enduring 90 minutes; Group size between 8-10 participants;
  Arms: Stepped and Collaborative Care Modell
Behavioral: Adolescent-Groupintervention — Target group: Adolescent participants with moderate depressive symptoms. Therapists: Two child and adolescent psychiatrists with translators or two native speaking child and adolescent psychotherapists.
  Content: Elements which are based on the START-Manual13 teaching emotion recognition and emotion regulation; Foundations are based on Dialetical behavior therapy; Specific focus lies on the use of mindfulness; Additionally the social network of the participants will receive psycho-education; Professional helpers in facilities will acquire E-learning elements of the SHELTER-program (Safety and Help for Early Adverse Life events and Traumatic Experiences in minor refugees)
  Arms: Stepped and Collaborative Care Modell
Other: Treatment as Ususal — Participants will receive the currently conducted routine and standard psychiatric health care. This involves ambulatory and stationary treatment by board certificated psychiatrists and psychotherapists.
  Arms: Treatment as Usual

SUMMARY:
The objective of this study is to investigate a stepped and collaborative care model (SCCM) for adolescent and adult refugees suffering from depression living in Germany.

DETAILED DESCRIPTION:
A prospective, cluster-randomized intervention study, conducted in seven German cities and comprising a total of 476 patients, should compare effectiveness and efficiency of this SCCM as compared to a 'Treatment as Usual' (TAU) condition. The fundamental principle of the examined care model is to provide patients with mild and moderate depression with accessible and affordable treatments, which are located outside the usual psychiatric-psychotherapeutic institutions (e.g. peer-to-peer-approaches or smartphone based interventions).

The acquired insights from the stepped care model, as well as concerning the individual low barrier interventions for adolescents and adults, can be used immediately for benefitting the provision of care of refugees but also for improving care of other communities with lacking access to health care systems. The generated disease figures from the nationwide screening process can be utilized directly to manage the provision of mental health fostering offers for refugees by federal institutions and social health insurance companies.

In both treatment arms (SCCM and TAU) and independent of intervention form participants will be assessed at four time periods after the initial screening process: Baseline (T1), after week 12 (T1), after week 24 (T2), after week 48 (T3).

Following clinical measurement tools will be used at all time periods:

* Refugee Health Screener (RHS-15)
* Patient Health Questionnaire (PHQ-9)
* Patient Health Questionnaire-Adapted (PHQ-A) *
* Montgomery-Åsberg Depression Scale (MÅDRS)
* Mannheimer Modul Ressourcenverbrauch (MRV)
* Brief Resilience Scale (BRS)
* General Self-Efficacy Scale (GSE)
* World Health Organization Quality of Life (WHOQOL-BREF)
* Child & Adolescent Trauma Screening (CATS)*

Following clinical measurement tools will be used at Baseline (T1):

* Demographics / Migration Questionnaires
* M.I.N.I. International Neuropsychiatric Interview
* M.I.N.I. KID International Neuropsychiatric Interview*
* Harvard Trauma Questionnaire (HTQ)

Following clinical measurement tools will be used at Baseline (T0) and after Post-Intervention (T1):

* Cultural Differences Subscale
* Credibility / Expectancy Questionnaire

Following clinical measurement tools will be used at Baseline (T0), after Post-Intervention (T1) and Follow-Up 1 (T3):

- Strengths and Difficulties Questionnaire (SDQ)

*Adolescents only

ELIGIBILITY:
Inclusion Criteria:

* Obtained a statutory health insurance
* Approved residence status as a refugee, asylum seeker or asylee
* Mother tongue in Arabic or Farsi/Urdu or speaks English or German fluently
* Age between 16-65 years
* Participants shows relevant depressive symptoms measured by the PHQ-9 or PHQ-A

Exclusion Criteria:

* An existing schizophrenia or degenerative disorder
* Missing informed consent
* Possible suicidality
* Uncertain residence status

Ages: 14 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 584 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2020-03-01 (Actual)

PRIMARY OUTCOMES:
Depression severity measured by the Patient Health Questionnaire - 9 (PHQ-9) | Baseline,12, 24 and 48 weeks after randomization
  Significant reduction in depression severity as measured by the Patient Health Questionnaire - 9 (PHQ-9) from baseline to post intervention in the experimental condition (SCCM) compared to the active control condition (TAU)

SECONDARY OUTCOMES:
Response and remission rates measured by the Mannheimer Modul Ressourcenverbrauch (MRV) | Baseline, 12, 24 and 48 weeks after randomization
  Exploreing the superiority of broader effectiveness parameters, such as response and remission rates measured by the MRV between the SCCM and TAU condition.
Traumatic events measured by the Child and Adoleszent Trauma Screening (CATS) | Baseline, 12, 24 and 48 weeks after randomization
  Significant reduction in emotional stress experienced by traumatic experiences as measured by the Child and Adoleszent Trauma Screening (CATS) in adolescents refugees from baseline to post intervention in the experimental condition (SCCM) compared to the active control condition (TAU)

CONTACTS AND LOCATIONS:
Overall Officials: Malek Bajbouj, Prof. Dr. med., Principal Investigator — Charite University, Berlin, Germany
Locations (1):
- Central Institute of Mental Health, Mannheim, Germany

REFERENCES:
- [Derived] Strupf M, Hoell A, Bajbouj M, Boge K, Wiechers M, Karnouk C, Kamp-Becker I, Banaschewski T, Meyer-Lindenberg A, Rapp M, Hasan A, Falkai P, Habel U, Heinz A, Plener P, Kaiser F, Weigold S, Mehran N, Ubleis A, Padberg F. Shared sorrow, shared costs: cost-effectiveness analysis of the Empowerment group therapy approach to treat affective disorders in refugee populations. BJPsych Open. 2023 Jun 22;9(4):e113. doi: 10.1192/bjo.2023.504. PMID 37345544
- [Derived] Boge K, Karnouk C, Hoell A, Tschorn M, Kamp-Becker I, Padberg F, Ubleis A, Hasan A, Falkai P, Salize HJ, Meyer-Lindenberg A, Banaschewski T, Schneider F, Habel U, Plener P, Hahn E, Wiechers M, Strupf M, Jobst A, Millenet S, Hoehne E, Sukale T, Dinauer R, Schuster M, Mehran N, Kaiser F, Brocheler S, Lieb K, Heinz A, Rapp M, Bajbouj M. Effectiveness and cost-effectiveness for the treatment of depressive symptoms in refugees and asylum seekers: A multi-centred randomized controlled trial. Lancet Reg Health Eur. 2022 Jun 6;19:100413. doi: 10.1016/j.lanepe.2022.100413. eCollection 2022 Aug. PMID 35694653